CLINICAL TRIAL: NCT04589572
Title: Structural and Funcional Outcomes of Extreme Lateral Interbody Fusion (XLIF) Compared to Posterior Lumbar Interbody Fusion (PLIF)
Brief Title: Extreme Lateral Interbody FusionFUSION (XLIF) Versus Posterior Lumbar Interbody Fusion (PLIF)
Acronym: XLIF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID-19
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Sint-Trudo Hospital (Other); Sint-Franciscus Ziekenhuis (Unknown)
Responsible Party: Principal Investigator, Frank Vandenabeele, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UH-XLIF-001
Record Dates: First submitted 2020-07-16; First posted 2020-10-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Muscle Damage; Atrophy; Degenerative Diseases, Spinal Cord
MeSH Terms: conditions — Atrophy; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: EXTREME LATERAL INTERBODY FUSION (XLIF) VERSUS POSTERIOR LUMBAR INTERBODY FUSION (PLIF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XLIF - group (Experimental)
  Interventions: Procedure: XLIF
- PLIF - Group (Active Comparator)
  Interventions: Procedure: PLIF

INTERVENTIONS:
Procedure: XLIF — the XLIF procedure, a minimally invasive procedure that approaches the spine from the lateral via the space between the 12th rib and the highest point of the iliac crest.
  Arms: XLIF - group
Procedure: PLIF — open posterior lumbar interbody fusion (PLIF) or transforaminal lumbar interbody fusion (TLIF) are used to treat degenerative diseases of the spinal column.
  Arms: PLIF - Group

SUMMARY:
Since the first successful spinal fusion surgery using a modern stabilization technique in 1909, surgical fusion has become one of the most commonly performed procedures for degenerative disease of the lumbar spine. The incidence of lumbar spinal fusion for degenerative conditions has more than doubled from 2000 until 2009. Despite the high incidence of fusion surgery, the decision making in lumbar fusion surgery is complicated by a wide variety of indications (the greatest measured in any surgical procedure). This could indicate there might be an overuse of lumbar fusion. However, decompression alone, or non-operative care for degenerative conditions may risk progressive spinal instability, intractable pain, and neurological impairment. These complications in the absence of fusion surgery, clearly demonstrate the beneficial effects of adding spinal fusion surgery. Because of its beneficial effect and high usage, it is of greatest importance to reduce postoperative disability and pain, by diminishing surgical invasiveness.

Traditional open posterior lumbar interbody fusion (PLIF) or transforaminal lumbar interbody fusion (TLIF) are used to treat degenerative diseases of the spinal column. These techniques require an extensive dissection of the paraspinal musculature, which in term can lead to muscle denervation, loss of function, muscular atrophy, and spinal instability. It has also been known that paraspinal muscle damage induced during surgery is related to long term disability and pain. With this knowledge, minimally invasive spine surgery began to develop in the mid-twentieth century. Since then, new direct approaches to the lumbar spine, known as lumbar lateral interbody fusion (LLIF), direct lateral interbody fusion (DLIF), or extreme lateral interbody fusion (XLIF), have been introduced.

This study will focus on XLIF. Ozgur. 2006 first reported the XLIF procedure, as a minimally invasive procedure that approaches the spine from the lateral via the space between the 12th rib and the highest point of the iliac crest. This approach allows direct access to the intervertebral disc space without disruption of the peritoneal structures or posterior paraspinal musculature. Ohba. 2017 compared XLIF with percutaneous pedicle screws to traditional PLIF, and found that PLIF was associated with less intraoperative blood loss, postoperative white blood cell (WBC) counts, C-reactive protein (CRP) levels, and creatine kinases (CK) levels, indicating less muscle damage. Postoperative recovery of performance was significantly faster in the XLIF group. 1-year disability and pain scores were also significantly lower in the XLIF group. Despite these significant better results reported in the XLIF group, the systematic review of Barbagallo. 2015 concluded that there is insufficient evidence of the comparative effectiveness of lateral lumbar interbody fusion (XLIF) versus PLIF/ TLIF surgery. This indicates that the evidence for choosing between XLIF or a traditional approach is still scarce, and no recommendations can be made.

This study will focus on comparing XLIF to PLIF. The objective of this study is to compare clinical and structural outcome measures between the XLIF and PLIF groups, to confirm our hypothesis that the minimally invasiveness of the XLIF technique facilitates a significant faster post-operative recovery, and improves functional and structural outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical single level disc degeneration
* Age between 18 and 65 years old
* Understand Dutch (writing and speaking)
* Symptom duration ≤ 5 years

Exclusion Criteria:

* Involvement of the L5-S1 or L2-L3 segment
* Psychiatric pathology/ problems (e.g. substance abuse)
* Pregnancy
* Being non-suitable for surgery
* BMI ≥35
* Other diagnosed neurological or musculoskeletal diseases that might affect the spinal column
* Not being able to function independently (activities of daily living)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Paraspinal muscle biopsy | - 1 week
  From each participant a sample will be obtained from the lumbar multifidus and erector spinae muscle before (T0) and after lumbar surgery (T4). These samples will be obtained using a minimally invasive ultrasound guided percutaneous biopsy technique using a local anesthetic. The samples will be immediately frozen. After cutting these will be used for immunofluorescent staining for myosin heavy chain I, IIA, and IIX. These staining's will be analyzed to measure muscle fiber size and number. These data will be used to evaluate within and between group differences in atrophy or shift in muscle fiber typing.
Paraspinal muscle biopsy | week 8
  From each participant a sample will be obtained from the lumbar multifidus and erector spinae muscle before (T0) and after lumbar surgery (T4). These samples will be obtained using a minimally invasive ultrasound guided percutaneous biopsy technique using a local anesthetic. The samples will be immediately frozen. After cutting these will be used for immunofluorescent staining for myosin heavy chain I, IIA, and IIX. These staining's will be analyzed to measure muscle fiber size and number. These data will be used to evaluate within and between group differences in atrophy or shift in muscle fiber typing.
concentration of C-Reactive Protein | - 1 week
  Blood analysis
concentration of C-Reactive Protein | 24 hours after surgery
  Blood analysis
concentration of C-Reactive Protein | 48 hours after surgery
  Blood analysis
concentration of C-Reactive Protein | week 8
  Blood analysis
concentration of Calcium | - 1 week
  Blood analysis
concentration of Calcium | 24 hours after surgery
  Blood analysis
concentration of Calcium | 48 hours after surgery
  Blood analysis
concentration of Calcium | week 8
  Blood analysis
concentration of Phosphate | - 1 week
  Blood analysis
concentration of Phosphate | 24 hours after surgery
  Blood analysis
concentration of Phosphate | 48 hours after surgery
  Blood analysis
concentration of Phosphate | week 8
  Blood analysis
concentration of Creatine kinase | - 1 week
  Blood analysis
concentration of Creatine kinase | 24 hours after surgery
  Blood analysis
concentration of Creatine kinase | 48 hours after surgery
  Blood analysis
concentration of Creatine kinase | week 8
  Blood analysis
concentration of Myoglobine | - 1 week
  Blood analysis
concentration of Myoglobine | 24 hours after surgery
  Blood analysis
concentration of Myoglobine | 48 hours after surgery
  Blood analysis
concentration of Myoglobine | week 8
  Blood analysis
concentration of Lactate dehydrogenase | - 1 week
  Blood analysis
concentration of Lactate dehydrogenase | 24 hours after surgery
  Blood analysis
concentration of Lactate dehydrogenase | 48 hours after surgery
  Blood analysis
concentration of Lactate dehydrogenase | week 8
  Blood analysis
concentration of Alkaline phosphatase | - 1 week
  Blood analysis
concentration of Alkaline phosphatase | 24 hours after surgery
  Blood analysis
concentration of Alkaline phosphatase | 48 hours after surgery
  Blood analysis
concentration of Alkaline phosphatase | week 8
  Blood analysis

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | - 1 week
  MRI images will be used to evaluate paraspinal and iliopsoas muscle cross-sectional area (CSA), and functional cross-sectional area (FCSA).
Magnetic Resonance Imaging (MRI) | week 8
  MRI images will be used to evaluate paraspinal and iliopsoas muscle cross-sectional area (CSA), and functional cross-sectional area (FCSA).
DEXA-san (Dual-energy X-ray Absorptiometry). | - 1 week
  Participants will undergo a DEXA-scan to evaluate body composition
DEXA-san (Dual-energy X-ray Absorptiometry). | week 8
  Participants will undergo a DEXA-scan to evaluate body composition
activity tracker | From - 1 week up to week 8 (24 hours a day)
  Participant will were an activity tracker from -1 week -1 until week 8 to compare activity patterns between groups
Visual analogue scale (VAS) | - 1 week
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Visual analogue scale (VAS) | 24 hours after surgery
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Visual analogue scale (VAS) | 48 hours after surgery
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Visual analogue scale (VAS) | week 8
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Pain catastrophizing scale (PCS) | - 1 Week
  Participants are asked to indicate the degree to which they have specific thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale.
Pain catastrophizing scale (PCS) | week 8
  Participants are asked to indicate the degree to which they have specific thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale.
Pain vigilance and awareness questionnaire (PVAQ) | - 1 week
  The PVAQ is a 16-item measure of attention to pain that assesses awareness, consciousness, vigilance, and observation of pain.
Pain vigilance and awareness questionnaire (PVAQ) | week 8
  The PVAQ is a 16-item measure of attention to pain that assesses awareness, consciousness, vigilance, and observation of pain.
Oswestry Disability Index (ODI) | - 1 week
  This is a questionnaire than has been proven valid and reliable to evaluate the restrictions that people with low back pain experience during their daily living. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Oswestry Disability Index (ODI) | week 8
  This is a questionnaire than has been proven valid and reliable to evaluate the restrictions that people with low back pain experience during their daily living. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
EQ5D questionaire | - 1 week
  The EQ-5D is a standardized questionnaire in which five levels of health (mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression ) can be scored. The patients also has to indicate how he/she experiences their health state on a scale from 0 to 100.
EQ5D questionaire | week 8
  The EQ-5D is a standardized questionnaire in which five levels of health (mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression ) can be scored. The patients also has to indicate how he/she experiences their health state on a scale from 0 to 100.
Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) | - 1 week
  The PASIPD is a reliable and valid questionnaire consisting of 13 items to measure the physical activity of people with disabilities. The average hours per day for each item is scored, and is multiplied by a metabolic equivalent (MET) value associated with the intensity of the activity and summing over items 2 through 13. Scores range from 0 (no activity) to >100 METS hour/day (very high).
Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) | week 8
  The PASIPD is a reliable and valid questionnaire consisting of 13 items to measure the physical activity of people with disabilities. The average hours per day for each item is scored, and is multiplied by a metabolic equivalent (MET) value associated with the intensity of the activity and summing over items 2 through 13. Scores range from 0 (no activity) to >100 METS hour/day (very high).
The Tampa Scale for Kinesiophobia (TSK) | - 1 week
  : The TSK is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. The higher the score the more fear of movement will be present, with a maximum score of 68. The cut of value to state a patient is experiencing fear of movement is 37/68.
The Tampa Scale for Kinesiophobia (TSK) | week 8
  : The TSK is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. The higher the score the more fear of movement will be present, with a maximum score of 68. The cut of value to state a patient is experiencing fear of movement is 37/68.
The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | - 1 week
  The PS is a simple measure of functional status, originally developed by the ECOG to evaluate cancer treatment toxicity. It has scores from 0-5 that correlate with the Karnofsky scale. Although this instrument has been developed to evaluate cancer treatment, it has been used to evaluate the post-operative performance status in persons undergoing lumbar surgery
The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | 24 hours after surgery
  The PS is a simple measure of functional status, originally developed by the ECOG to evaluate cancer treatment toxicity. It has scores from 0-5 that correlate with the Karnofsky scale. Although this instrument has been developed to evaluate cancer treatment, it has been used to evaluate the post-operative performance status in persons undergoing lumbar surgery
The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | 48 hours after surgery
  The PS is a simple measure of functional status, originally developed by the ECOG to evaluate cancer treatment toxicity. It has scores from 0-5 that correlate with the Karnofsky scale. Although this instrument has been developed to evaluate cancer treatment, it has been used to evaluate the post-operative performance status in persons undergoing lumbar surgery
The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | week 8
  The PS is a simple measure of functional status, originally developed by the ECOG to evaluate cancer treatment toxicity. It has scores from 0-5 that correlate with the Karnofsky scale. Although this instrument has been developed to evaluate cancer treatment, it has been used to evaluate the post-operative performance status in persons undergoing lumbar surgery
Dietary intake | up to week 8
  Participant will be asked to register their food intake using a standardized form. This will be done on two week days, and one day during the weekend. This outcome will be used to asses a difference in protein intake, that might affect muscle atrophy after surgery (control parameter).
Blood loss | week o
  Surgical blood loss needs to be reported in milliliters.
Operating time | week o
  Time from the incision until closing of the operating site will be reported.
Complications | week o
  Bleeding, infection, nerve damage, re-intervention, permanent injuries will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandenabeele, prof. dr., Principal Investigator — Hasselt University; Sjoerd stevens, drs., Study Chair — Hasselt University
Locations (3):
- Belgium (3):
  - Jessa Ziekenhuis, Hasselt
  - Sint-Franciscus Ziekenhuis, Heusden-Zolder
  - Sint-Trudo Ziekenhuis, Sint-Truiden